CLINICAL TRIAL: NCT02215980
Title: A PHASE III, MULTICENTRE, RANDOMIZED, CONTROLLED STUDY TO DETERMINE THE EFFICACY AND SAFETY OF STANDARD SCHEDULE VERSUS A NEW ALGORITHM OF DOSE REDUCTIONS IN ELDERLY AND UNFIT NEWLY DIAGNOSED MULTIPLE MYELOMA PATIENTS RECEIVING LENALIDOMIDE PLUS STEROIDS
Brief Title: STUDY TO DETERMINE THE EFFICACY AND SAFETY OF STANDARD SCHEDULE VERSUS A NEW ALGORITHM OF DOSE REDUCTIONS IN ELDERLY AND UNFIT NEWLY DIAGNOSED MULTIPLE MYELOMA PATIENTS RECEIVING LENALIDOMIDE PLUS STEROIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-PI-0752
Record Dates: First submitted 2014-07-28; First posted 2014-08-13 (Estimated); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Diagnosis; Elderly and unfit patients; Lenalidomide plus steroids
MeSH Terms: conditions — Multiple Myeloma; Disease | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): * Lenalidomide: at the dose of 25 mg/daily as oral administration (PO) on days 1-21.
  * Dexamethasone: at the dose of 20 mg as oral administration (PO) once weekly. Each cycle will be repeated every 28 days until progression or intolerance.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone
- B (Experimental): * Lenalidomide: at the dose of 25 mg/daily as oral administration (PO) on days 1-21
  * Dexamethasone: at the dose of 20 mg as oral administration (PO) once weekly. Each cycle will be repeated every 28 days, for a total of 9 cycles.
  Maintenance until progression or intolerance:
  - Lenalidomide: 10 mg/daily on days 1-21 of each 28-day cycle
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide
Drug: Dexamethasone

SUMMARY:
This protocol is a phase III multicenter, randomized, controlled study designed to assess the safety and the efficacy of standard schedule versus a new algoritm of dose reductions in elderly and unfit newly diagnosed Multiple Myeloma (MM) patients receiving lenalidomide plus steroids.

DETAILED DESCRIPTION:
TREATMENT PERIOD:

Arm A: Rd

* Lenalidomide: at the dose of 25 mg/daily as oral administration (PO) on days 1-21.
* Dexamethasone: at the dose of 20 mg as oral administration (PO) once weekly. Each cycle will be repeated every 28 days until progression or intolerance.

Arm B: Rd-R (reduced)

* Lenalidomide: at the dose of 25 mg/daily as oral administration (PO) on days 1-21
* Dexamethasone: at the dose of 20 mg as oral administration (PO) once weekly. Each cycle will be repeated every 28 days, for a total of 9 cycles.

Maintenance until progression or intolerance:

- Lenalidomide: 10 mg/daily on days 1-21 of each 28-day cycle

ELIGIBILITY:
Inclusion Criteria:

* Patients >65 years unfit and unsuitable, according to the investigator's opinion, to receive approved first line treatments for newly diagnosed MM.
* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Symptomatic MM based on standard CRAB criteria (5).
* Patient has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, ≥ 0.5 g/dL of M-protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours. For patients with oligo or non-secretory MM, it is required that they have measurable plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan) or an abnormal free light chain ratio (n.v.: 0.26-1.65). We anticipate that less than 10% of patients admitted to this study will be oligo- or non-secretory MM with free light chains only in order to maximize interpretation of benefit results.
* All randomized patients will be selected based on the use of 3 geriatric scales: IADL, ADL, Charlson. Unfit patients with clinical sign of frailty (mild, moderate or severe frailty), including need help for household tasks and personal care can be enrolled in this trial (2,4).
* In order to include patients who normally are not select for clinical trials, also patients with the following abnormal laboratory values can be considered:

  1. absolute neutrophil count (ANC) < 1 x 10^9/L
  2. platelet count < 80 x 10^9/L
  3. haemoglobin < 8 g/dl.
  4. aspartate transaminase (AST): < 5 x the upper limit of normal (ULN).
  5. alanine transaminase (ALT): < 5 x the ULN.
  6. total bilirubin: > 1.5 x the ULN
  7. calculated or measured creatinine clearance: <30 mL/minute

The geriatric assessment evaluations will select unfit patients to be randomized regardless of possible abnormal laboratory values at the study entry.

Exclusion Criteria:

* Pregnant or lactating females.
* Male patients not agreeing to use an acceptable method for contraception (i.e., condom or abstinence) for the duration of the study.
* Females of childbearing potential not agreeing to use two acceptable methods for contraception (e.g. a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid < to the equivalent of dexamethasone 40 mg/day for 4 days).
* Any significant medical disease or conditions that, in the investigator's opinion, may interfere with protocol adherence or subject's ability to give informed consent or could place the subject at unacceptable risk.
* Presence of clinical active infectious hepatitis type B or C, classified into Child-Pugh class C (see Appendix V) and HIV.
* Presence of acute active infection requiring antibiotics or infiltrative pulmonary disease.
* Contraindication to any of the required drugs or supportive treatments.
* Presence of prior history of malignancies, other than multiple myeloma, with a life expectancy < 2 years.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 3 years
  Determine the Event-free survival defined as:
  * Progression
  * Death for any cause
  * Discontinuation of lenalidomide therapy
  * Occurrence of any haematological grade 4 or non-haematological grade 3-4 adverse events (AES), including Secondary Primary Malignancies (SPMs)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 5 years
Overall survival (OS) | 5 years
Time to progression (TTP) | 5 years
Overall response rate (ORR) | 5 years
Time to response (TTR) | 5 years
Duration of response (DOR) | 5 years
Time to the next therapy (TNT) | 5 years
Incidence of dose reduction and drug discontinuation | 5 years
Health care cost | 5 years
Correlation between tumor response and outcome with baseline prognostic factors | 5 years
  Analysis of tumor response and outcome stratification by prognostic factors
Quality of life assessment (HRQOL) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione EMN Italy Onlus, Torino, Italy

REFERENCES:
- [Derived] Larocca A, Bonello F, Gaidano G, D'Agostino M, Offidani M, Cascavilla N, Capra A, Benevolo G, Tosi P, Galli M, Marasca R, Giuliani N, Bernardini A, Antonioli E, Rota-Scalabrini D, Cellini C, Pompa A, Monaco F, Patriarca F, Caravita di Toritto T, Corradini P, Tacchetti P, Boccadoro M, Bringhen S. Dose/schedule-adjusted Rd-R vs continuous Rd for elderly, intermediate-fit patients with newly diagnosed multiple myeloma. Blood. 2021 Jun 3;137(22):3027-3036. doi: 10.1182/blood.2020009507. PMID 33739404